CLINICAL TRIAL: NCT05891795
Title: Topical Androgen Receptor Inhibitor for Steroid-related Acne Vulgaris in Transgender Male Patients Receiving Masculinizing Hormone Therapy
Brief Title: Clascoterone for Steroid-related Acne Vulgaris in Transgender Male Patients Receiving Masculinizing Hormone Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anne Chang, Professor of Dermatology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69870
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking will occur by the investigational pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clascoterone (Experimental)
  Interventions: Drug: Clascoterone 1% Top Cream
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Clascoterone 1% Top Cream — Apply a thin layer to the affected area twice daily.
  Arms: Clascoterone
Drug: Vehicle — Apply a thin layer to the affected area twice daily.
  Arms: Vehicle

SUMMARY:
Mechanism-based acne treatment for transgender patients receiving testosterone currently does not exist and is an unmet medical need. This study explores clascoterone to treat testosterone induced acne. Many treatments we use to treat acne in females cannot be used in transgender males because they interfere with hormone therapy. Androgens have been associated with the development of acne vulgaris. Recently, a topical androgen receptor inhibitor cream (clascoterone) has been FDA-approved for the treatment of acne. However, clinical trials of clascoterone have excluded participants on exogenous hormones. Clascoterone has been hypothesized to be effective in the treatment of acne in transgender male participants on masculinizing hormone therapy, but it has never been studied or reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* transgender male or gender diverse patient on MHT
* on a stable dose of MHT for at least 3 months prior to the study
* anticipate being on the same dose of MHT for the duration of the study
* have steroid-related acne vulgaris as determined by the investigator with onset or worsening after initiation of MHT
* have at least 20 papules or pustules on the face
* consistent skin care regimen (topical and systemic medications) for at least 4 weeks prior to enrollment and continue it for the duration of the study (however, note exclusion below that topical steroids on face not allowed for 4 weeks prior to enrollment and during study)*;
* age 16 years old or older
* potential participants who have ovaries and are or planning to be sexually active with partners that produce sperm will need to use a medically reliable form of birth control (including but not limited to condoms, intrauterine device, oral contraceptives) before enrollment and during the study

  * Note inhaled steroids are allowed as long as regimen is stable one month prior to enrollment and during the study

Exclusion Criteria:

* changes in topical or systemic anti-acne medications or procedures within four weeks of study enrollment
* use of topical steroids on the face within 4 weeks prior to enrollment and during study
* pregnant or breast-feeding patients
* unable to provide informed consent, follow the protocol, attend study visits, or any other circumstance or condition which the investigator deems may obscure interpretation of results or affect safety of the potential participant.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of papules/pustules | Week 0, and week 12
  Total count of papules (including pustules) will be measured on the entire face at screening and monthly during the three month treatment period. Change in total papules count will be used to compare the efficacy of clascoterone 1% cream versus vehicle at time point week 12 versus week 0.

SECONDARY OUTCOMES:
Change in serum testosterone | Week 0, and week 12
  Serum testosterone will be measured before starting the treatment (week 0) and following the 3-month course (week 12). We will use the change in serum testosterone to investigate if clascoterone, a local androgen receptor inhibitor, has systemic effects for transgender patients on MHT.
Change in sebum output | Week 0, and week 12
  Sebum output will be measured using a Sebumeter SM815 probe (Courage & Khazaka, Köln or Cologne, Germany) before starting the treatment (week 0) and following the 3-month course (week 12). The specifications for the Sebumeter are as follows: Infrared 950 nanometers LED light, Type LED SFH 420 IR 950 nanometers, 1.8 voltz, 50 mAmps, CHIP-SMD. This specific apparatus has been used in several previous acne vulgaris studies. The patient will be asked to not use any topical preparations on their face 24 hours prior to these appointments. Measurements will be taken from the forehead.
Change in Acne-QoL and AI-ADL scores | Week 0, and week 12
  Patient reported outcomes will be measured using Acne-QoL and AI-ADL (only for participants 18+ years old) before starting the treatment (week 0) and following the 3-month course (week 12).
Change in microbiomic profile (measured by relative species abundance) | Week 0, and week 12
  Skin microbiome samples will be taken from the nose using noninvasive bacterial swab following the instructions of the manufacturer before starting the treatment (week 0) and following the 3 month course (week 12). Sample preparation and subsequent shotgun sequencing on microbiome samples will be done commercially (Microbiome Insights). Shotgun metagenomic sequencing will be performed using Illumina 2x150 paired-end reads with a mean read depth of at least 6-7 million sequences per sample. High quality reads will undergo taxonomic profiling to obtain relative abundances. Change in relative species percentage & abundance will be used as a correlate for treated versus placebo, responders versus non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lynn S Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No